CLINICAL TRIAL: NCT01843699
Title: Double-blind Placebo Controlled Topiramate Trial for Pathological Gamblers
Brief Title: Topiramate Trial for Pathological Gamblers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Hermano Tavares, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1341/06
Record Dates: First submitted 2013-04-23; First posted 2013-05-01 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Pathological Gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Topiramate (Experimental): A 12-week topiramate flexible dose administration plus 4 sessions of a manualized cognitive restructuring intervention.
  Interventions: Drug: Topiramate flexible dosage; Behavioral: 4-session gambling cognitive restructuring
- Placebo (Placebo Comparator): A 12-week placebo matching tablets plus 4 sessions of a manualized cognitive restructuring intervention.
  Interventions: Drug: Placebo matching tablets; Behavioral: 4-session gambling cognitive restructuring

INTERVENTIONS:
Drug: Topiramate flexible dosage
  Arms: Topiramate
Drug: Placebo matching tablets
  Arms: Placebo
Behavioral: 4-session gambling cognitive restructuring

SUMMARY:
Objectives: Pathological gambling (PG) is a prevalent disorder with no approved pharmacological treatment. Previous reports suggest that topiramate could be useful in reducing impulsivity in PG, and craving in other addictions. The goal of this study was to investigate the effectiveness of topiramate combined with brief cognitive restructuring in treating PG. Methods: 38 PG patients were randomized to either topiramate (N=18) or placebo (N=20) in a 12-week double-blind trial; all patients received brief cognitive restructuring. The main outcome measures were craving, gambling behaviour, gambling cognitive distortions, impulsivity, depression and social adjustment.

ELIGIBILITY:
Inclusion Criteria:

* current Diagnostic and Statistical Manual Fourth Edition Text Revised (DSM-IV-TR) diagnosis of pathological gambling
* a betting frequency of at least once a week in the last 30 days
* women within fertility age had to be already practicing an acceptable contraception method and to be negative at a pregnancy test.

Exclusion Criteria:

* illiteracy
* breastfeeding for women
* previous history of alcohol abuse/dependence with current elevation of liver enzymes, or a present diagnosis of alcohol abuse/dependence
* past or current drug abuse/dependence, except for nicotine dependence
* history of current or past DSM-IV-TR diagnosis of bipolar disorder, schizophrenia, psychosis or any neuropsychiatric condition causing cognitive impairment
* a history of suicide attempt or acute suicide risk
* severe depression indicated by a score equal to or higher than 30 at the Beck Depression Inventory
* current participation in psychotherapy for pathological gambling, including Gamblers Anonymous in the past 3 months
* current use of mood stabilizers, antidepressants, antipsychotics, except occasional use of benzodiazepines
* cardiovascular disease including a history of heart attack, stroke, arrhythmia, cardiac failure in the past 5 years
* chronic or acute renal and liver failure
* a personal or family history of nephrolithiasis
* immunodeficiency
* any blood dyscrasia.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Gambling craving | 12 weeks
  The scale selected for this purpose was The Gambling Symptom Assessment Scale (G-SAS), it is a one-dimension self-report scale which assesses mostly gambling craving, related thoughts and behaviors. Reference: Kim SW, Grant JE, Potenza MN, Blanco C, Hollander E. The Gambling Symptom Assessment Scale (G-SAS): a reliability and validity study. Psychiatry Res. 2009 Mar 31;166(1):76-84.

SECONDARY OUTCOMES:
Gambling behavior | 12 weeks
  Includes frequency of betting, amount of money and time spent on gambling over a month

OTHER OUTCOMES:
Social adjustment | 12 weeks
  The Social Adjustment Scale (SAS) is a self-report scale that assesses seven specific areas: work, social life and leisure, extended family relationship, marital relationship, relationship with offspring, domestic life and financial situation. References:
  1. Weissman MM, Bothwell S, (1976): Assessment of social adjustment by patient self-report. Arch Gen Psychiatry 33:1-5.
  2. Gorenstein C, Moreno RA, Bernick MA, Carvalho SC, Nicastri S, Cordas T, et al, (2002): Validation of the Portuguese version of the Social Adjustment Scale on Brazilian samples. Journal of Affective Disorders 69: 167-175.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Psiquiatria da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Dowling N, Merkouris S, Lubman D, Thomas S, Bowden-Jones H, Cowlishaw S. Pharmacological interventions for the treatment of disordered and problem gambling. Cochrane Database Syst Rev. 2022 Sep 22;9(9):CD008936. doi: 10.1002/14651858.CD008936.pub2. PMID 36130734